CLINICAL TRIAL: NCT04893642
Title: To Resect or Not Resect - The Randomized Swedish Rectal Prolapse Trial
Brief Title: Swedish Rectal Prolapse Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study had planned to recruit 220 but was termianted in advance when 134 patients were randomized. This was done due to slow recruitment.
Sponsor: Danderyd Hospital (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Klas Pekkari, Head of Colorectal unit, Senior consultant, Md, PhD, Danderyd Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: swedishrectalprolapse
Record Dates: First submitted 2021-04-27; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Rectal Prolapse
Keywords: Randomized controlled study; Multicenter; Prospective
MeSH Terms: conditions — Rectal Prolapse

STUDY DESIGN:
Intervention Model Description: This was a multicenter randomized trial with a 2 x 2 factorial design conducted in 13 sites in Sweden. Randomization was performed with randomly assigned envelopes, stratified for each participating center. Patients were randomized between perineal and abdominal approach (A). The perineal group was further randomized to Delorme's or Altemeier's procedure (B) and the abdominal group to suture rectopexy or resection rectopexy (C). Patients who were considered unsuitable for random allocation to a perineal or an abdominal procedure were included only in (B) or (C).
Who Masked: Outcomes Assessor
Masking Description: Masking was done for outcome assessor concerning the answers for questionnaires that were the primary endpoint. Masking of arms were not done concerning recurrence of rectal prolapse.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Abdominal suture rectopexy (Active Comparator): Patients were randomized first into either an abdominal or a perineal approach. The abdominal group was then further randomized to suture rectopexy or resection rectopexy.
  Interventions: Procedure: Suture rectopexy
- Abdominal resection rectopexy (Active Comparator): Patients were randomized first into either an abdominal or a perineal approach. The abdominal group was then further randomized to suture rectopexy or resection rectopexy.
  Interventions: Procedure: resection rectopexy
- Perineal Delorme (Active Comparator): Patients were randomized first into either an abdominal or a perineal approach. The perineal group was then further randomized to Delorme's operation or Altemeier's operation.
  Interventions: Procedure: Delorme's operation
- Perineal Altemeier (Active Comparator): Patients were randomized first into either an abdominal or a perineal approach. The perineal group was then further randomized to Delorme's operation or Altemeier's operation.
  Interventions: Procedure: Altemeier's operation

INTERVENTIONS:
Procedure: Suture rectopexy
  Arms: Abdominal suture rectopexy
Procedure: resection rectopexy
  Arms: Abdominal resection rectopexy
Procedure: Delorme's operation
  Arms: Perineal Delorme
Procedure: Altemeier's operation
  Arms: Perineal Altemeier

SUMMARY:
Rectal prolapse is a medical condition where rectum is protruding through the anal opening. The treatment is by surgery that can be performed with an anterior approach through the abdomen or a posterior perineal approach. The condition is more common in elderly patients and much more common in women compared to men. All used surgical techniques have advantages and disadvantages. The primary aim of this study is to evaluate if an abdominal or perineal surgical approach is best to correct a rectal prolapse. The outcome measures will be validated questionnaires on quality of Life (SF-36) and bowel function (modified Wexner incontinence score) as well as recurrence of the rectal prolapse and surgical complications.

The study is a randomized multicenter trial with a 2x2 factorial design. Patients will be randomized between perineal and abdominal approach in a first randomization and the perineal group will then further be randomized into one of two specific operations (delorme or altemeier) and the abdominal group will be further randomized into suture rectopexy or resection rectopexy.

The patients will be followed for 3 months, 1 year and 3 years and a longterm follow up of up to 17 years for recurrence.

DETAILED DESCRIPTION:
Background Full thickness rectal prolapse, or procidentia, is a benign but distressing condition. It is defined as the circumferential protrusion of all layers of the rectal wall through the anal sphincters. The annual incidence is 2,5 per 100 000, predominantly in the elderly, and male-to-female ratio is about 1:6.

More than 100 different procedures have been described for surgical treatment of rectal prolapse and consensus has not yet been reached. Traditionally, perineal procedures have been reserved for older patients who are not fit for an abdominal operation. The two most common perineal procedures are Delorme's operation, i.e. mucosectomy and rectal plication, and perineal rectosigmoidectomy, also known as Altemeier's operation, which is a full-thickness excision of the rectum.

The choices between abdominal vs. perineal approach and resection or not were all addressed in the Swedish rectal prolapse trial with possible differences in bowel function, quality of life, recurrence rate and complications as end points.

Study design and randomization This was a multicenter randomized trial with a 2 x 2 factorial design conducted in 13 sites in Sweden. At inclusion, patients signed an informed consent form and the attending surgeon contacted the central trial office at the Danderyd Hospital, Stockholm, Sweden. Randomization was performed with randomly assigned envelopes, stratified for each participating center. Patients were randomized between perineal and abdominal approach (A). The perineal group was further randomized to Delorme's or Altemeier's procedure (B) and the abdominal group to suture rectopexy or resection rectopexy (C). Patients who were considered unsuitable for random allocation to a perineal or an abdominal procedure were included only in (B) or (C).

Preoperative evaluation and procedures All patients were clinically examined and diagnosed with full thickness rectal prolapse. Further examinations with endoscopy, colon transit studies, anorectal manometry, defecography, endoanal ultrasound and pudendal nerve motor latency were optional and were performed as indicated at each surgeon's discretion. Operative procedures were described in the study protocol, see appendix. Abdominal procedures were performed laparoscopically or as open procedure.

In order to validate data all questionnaires were gathered at the central trial hospital and inspected by a second researcher.

The surgical procedures were identified and standardized to a large extent. Both minimal invasive and open surgery were allowed. For example the abdominal procedures were described that mobilization of rectum should be done in the posterior aspect, the lateral ligaments should not be divided, Suture rectopexy should be done with non-absorbable 0.0 sutures, the cul de sac should not be closed.

The sample size was calculated to 220 patients in the first randomization between abdominal and perineal approach. With 220 patients a difference in recurrence of 13% could be identified with 90% power in a significance level of 5%. The plan was to analyze the categorical variables with either Fisher´s exact test or multivariate analysis.

A main study office was situated at Danderyd Hospital and randomization was done from this office at the time when the patient was scheduled for surgery. All hospitals performing surgery for rectal prolapses in Sweden were invited to the study.

ELIGIBILITY:
Inclusion Criteria:

1. Complete rectal prolapse
2. Informed consent
3. Surgical correction is considered appropriate
4. Capable to participate in follow-up visits and answering questionnaires

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2000-03-23 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Bowel function | 3 months
  Wexner incontinence score, points, 0-20, higher worse result
Bowel function | 1 year
  Wexner incontinence score, points, 0-20, higher worse result
Bowel function | 3 years
  Wexner incontinence score, points, 0-20, higher worse result
Quality of Life | 3 months
  SF-36, points, 0-100 points, higher better result
Quality of Life | 1 year
  SF-36, points, 0-100 points, higher better result
Quality of Life | 3 years
  SF-36, points, 0-100 points, higher better result

SECONDARY OUTCOMES:
Recurrence of rectal prolapse | 3 months
  recurrence at outpatient visits
Recurrence of rectal prolapse | 1 year
  recurrence at outpatient visits
Recurrence of rectal prolapse | 3 years
  recurrence at outpatient visits
Recurrence of rectal prolapse | through study completion, an average of 12 years
  Recurrence in Medical records

OTHER OUTCOMES:
Length of staý | up to 30 days after surgical intervention
  days
Blood loss at operation | during the surgical procedure
  milliliter
perioperative complications | up to 30 days after surgical intervention
  number classified by Clavien-Dindo

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Hjern, Ass Prof, MD, Principal Investigator — Danderyd Hospital; Klas Pekkari, Md PhD, Study Director — Danderyd Hospital
Locations (12):
- Sweden (12):
  - Sahlgrenska University Hospital, Gothenburg
  - Karlstad Central Hospital, Karlstad
  - Linköping University Hospital, Linköping
  - Sunderbyn Hopsital, Luleå
  - Skåne University Hospital, Malmo
  - Vrinnevi Hospital, Norrköping
  - Danderyd Hospital, Stockholm
  - karolinska Univeristy Hospital Solna, Stockholm
  - Karolinska University Hospital Huddiinge, Stockholm
  - Sankt göran hospital, Stockholm
  - Uddevalla Hospital, Uddevalla
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tou S, Brown SR, Nelson RL. Surgery for complete (full-thickness) rectal prolapse in adults. Cochrane Database Syst Rev. 2015 Nov 24;2015(11):CD001758. doi: 10.1002/14651858.CD001758.pub3. PMID 26599079
- [Background] Kairaluoma MV, Kellokumpu IH. Epidemiologic aspects of complete rectal prolapse. Scand J Surg. 2005;94(3):207-10. doi: 10.1177/145749690509400306. PMID 16259169
- [Background] Madiba TE, Baig MK, Wexner SD. Surgical management of rectal prolapse. Arch Surg. 2005 Jan;140(1):63-73. doi: 10.1001/archsurg.140.1.63. PMID 15655208
- [Background] Lundby L, Iversen LH, Buntzen S, Wara P, Hoyer K, Laurberg S. Bowel function after laparoscopic posterior sutured rectopexy versus ventral mesh rectopexy for rectal prolapse: a double-blind, randomised single-centre study. Lancet Gastroenterol Hepatol. 2016 Dec;1(4):291-297. doi: 10.1016/S2468-1253(16)30085-1. Epub 2016 Oct 4. PMID 28404199
- [Background] Senapati A, Gray RG, Middleton LJ, Harding J, Hills RK, Armitage NC, Buckley L, Northover JM; PROSPER Collaborative Group. PROSPER: a randomised comparison of surgical treatments for rectal prolapse. Colorectal Dis. 2013 Jul;15(7):858-68. doi: 10.1111/codi.12177. PMID 23461778
- [Background] Orwelius L, Nilsson M, Nilsson E, Wenemark M, Walfridsson U, Lundstrom M, Taft C, Palaszewski B, Kristenson M. The Swedish RAND-36 Health Survey - reliability and responsiveness assessed in patient populations using Svensson's method for paired ordinal data. J Patient Rep Outcomes. 2017;2(1):4. doi: 10.1186/s41687-018-0030-0. Epub 2018 Feb 7. PMID 29757320
- [Derived] Smedberg J, Graf W, Pekkari K, Hjern F. Comparison of four surgical approaches for rectal prolapse: multicentre randomized clinical trial. BJS Open. 2022 Jan 6;6(1):zrab140. doi: 10.1093/bjsopen/zrab140. PMID 35045155